CLINICAL TRIAL: NCT00034437
Title: Measurement of Cytomegalovirus (CMV)-Specific T Lymphocytes in CMV-Seropositive Normal Volunteers.
Brief Title: Immune Response to Cytomegalovirus
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020189; 02-H-0189
Record Dates: First submitted 2002-04-27; First posted 2002-04-29 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-04

CONDITIONS: Cytomegalovirus Infections
Keywords: Normal Volunteer; Phlebotomy; Cytomegalovirus; CMV; CMV Seropositve
MeSH Terms: conditions — Cytomegalovirus Infections

SUMMARY:
This study will evaluate immune responses against cytomegalovirus (CMV). About 80 percent of adults have been exposed to this virus. CMV typically remains dormant (inactive) in the body, causing no problems. In people with immune suppression, however, the virus can become reactivated and cause life-threatening pneumonia. The knowledge gained from this study may be useful in developing ways to improve immune responses to CMV in stem cell transplant recipients.

Healthy normal volunteers between 18 and 65 years of age who have been exposed to cytomegalovirus are eligible for this study. Candidates will be screened with a medical history and blood tests. Those enrolled will provide a 30-milliliter (6-tablespoon) blood sample once a week for 4 weeks and a final sample 2 months later. The blood will be used to design a test to detect immune responses against CMV and determine the differences in these responses among healthy individuals.

DETAILED DESCRIPTION:
The NHLBI Stem Cell Allotransplantation Program is researching methods to improve immunity against infectious organisms following allogeneic stem cell transplantation (SCT). We are particularly interested in cytomegalovirus (CMV), which can cause serious problems in patients following transplantation. In the future, we hope to design ways to improve immune responses to CMV in transplant recipients, such as vaccinating transplant donors and/or patients against this virus. In order to characterize the effect of any such intervention on CMV immunity, we first need to better understand CMV immune responses in normal, healthy persons. This involves designing and validating an in vitro assay, which can reliably and consistently detect immune responses against CMV. Furthermore, we hope to define the temporal variability that exists in CMV responses in healthy individuals, which is essential for the design and implementation of all future studies. We plan to collect blood samples from 20 normal volunteers who have been previously exposed to CMV (CMV seropositive individuals). Eligible individuals will be asked to donate blood on five occasions, once a week for four weeks and a fifth time, two months later. Eligible individuals must be 18-65 years of age, otherwise healthy, and seropositive for CMV exposure.

ELIGIBILITY:
INCLUSION CRITERIA:

Age 18-65

CMV seropositive

Informed consent given

EXCLUSION CRITERIA:

CMV seronegative

Abnormal blood counts (hemoglobin less than 12 g/dl, platelets less than 150,000/ul, absolute neutrophil count less than 1,500/ul, absolute lymphocyte count less than 1,000/ul)

Known history of heart, lung, kidney, liver, or bleeding disorder

Diagnosis of HIV infection

Diagnosis or suspicion of immunodeficiency state

History of intravenous drug use

Currently pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2002-04; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States